CLINICAL TRIAL: NCT06914674
Title: Tamoxifen for Advanced Solid Pseudopapillary Tumor of the Pancreas
Acronym: SPTP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Prof., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-14
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Neoplasms
Keywords: Solid Pseudopapillary Tumor of the Pancreas; Malignant; Advanced; Recurrence; Metastasis
MeSH Terms: conditions — Pancreatic Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: • Tamoxifen: 10 mg orally twice daily.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tamoxifen (Experimental): Tamoxifen: 10 mg orally twice daily. Combination therapy: Chemotherapy, radiotherapy, surgery, or other treatments per NCCN guidelines and patient condition.
  Interventions: Drug: Tamoxifen 20 mg

INTERVENTIONS:
Drug: Tamoxifen 20 mg — Tamoxifen: 10 mg orally twice daily. Combination therapy: Chemotherapy, radiotherapy, surgery, or other treatments per NCCN guidelines and patient condition.

SUMMARY:
Tamoxifen for Solid Pseudopapillary Tumor of the Pancreas

DETAILED DESCRIPTION:
Solid pseudopapillary tumor of the pancreas (SPTP) is a rare neoplasm, predominantly affecting young females, with unclear pathogenesis and hormonal receptor (estrogen/progesterone receptor) expression potentially influencing tumor behavior. While surgical resection is the standard treatment, patients with advanced, metastatic, or recurrent disease lack effective therapies. Case reports suggest tamoxifen, a selective estrogen receptor modulator, may improve outcomes in hormone receptor-positive SPTP. This trial aims to evaluate tamoxifen's efficacy and safety in advanced SPTP.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-80 years.
2. Histologically confirmed advanced SPTP with ER/PR+.
3. Advanced disease:

   * Unresectable primary tumor or distant metastasis (liver, lung, peritoneum, etc.).
   * Recurrent or refractory after prior surgery/systemic therapy.
4. ≥1 measurable lesion.
5. ECOG performance status 0-2.
6. Life expectancy ≥1 month.
7. Able to comply with study visits and oral medication.

Exclusion Criteria:

1. Non-SPTP pathology.
2. Active gastrointestinal inflammation/infection (e.g., pancreatitis).
3. Pregnancy/lactation.
4. Severe organ dysfunction (renal, cardiac, hepatic, or pulmonary).
5. Uncontrolled comorbidities (e.g., CNS disorders, unstable angina).
6. Conditions compromising patient safety or data integrity.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFSn) | 1 month
  Time from enrollment to disease progression

SECONDARY OUTCOMES:
Overall survival （OS） | 1 month
  OS of subjects from recruiting to the time of death from any cause
disease control rate (DCR) | 1 month
  disease control rate (DCR = CR + PR + SD)

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo Prof, MD, Principal Investigator — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kornietskaya A, Evdokimova S, Kachmazov A, Fedenko A, Bolotina L, Sidorov D, Volchenko N, Goeva N, Govaleshko A, Kaprin A. Endocrine therapy for metastatic solid pseudopapillary neoplasm of the pancreas: A case report. Front Oncol. 2022 Sep 13;12:970142. doi: 10.3389/fonc.2022.970142. eCollection 2022. PMID 36176411
- [Background] Guo M, Luo G, Jin K, Long J, Cheng H, Lu Y, Wang Z, Yang C, Xu J, Ni Q, Yu X, Liu C. Somatic Genetic Variation in Solid Pseudopapillary Tumor of the Pancreas by Whole Exome Sequencing. Int J Mol Sci. 2017 Jan 3;18(1):81. doi: 10.3390/ijms18010081. PMID 28054945
- [Background] Nishihara K, Tsuneyoshi M, Ohshima A, Yamaguchi K. Papillary cystic tumor of the pancreas. Is it a hormone-dependent neoplasm? Pathol Res Pract. 1993 Jun;189(5):521-6. doi: 10.1016/S0344-0338(11)80359-6. PMID 8378176
- [Background] Dominguez-Rosado I, Chan C, Ortiz-Hidalgo C, Chable-Montero F, Uscanga LF, Campuzano M, Robles-Diaz G. Immunohistochemical expression of luteinizing hormone receptor in solid pseudopapillary tumor of the pancreas. Pancreas. 2014 Aug;43(6):971-2. doi: 10.1097/MPA.0000000000000134. No abstract available. PMID 25010708